CLINICAL TRIAL: NCT01348945
Title: Proprioceptive Function, Postural Stability & Clinical Outcome After Stump Preserving Anterior Cruciate Ligament Reconstruction Surgery - A Comparative Study
Brief Title: Proprioceptive Function, Postural Stability & Clinical Outcome After Stump Preserving Anterior Cruciate Ligament Reconstruction Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Holly Leung King Ho, Physiotherapy Department of Prince of Wales Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SPACL-CS
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2010-12

CONDITIONS: Ruptured Anterior Cruciate Ligament; Partial Tear Ligament
Keywords: Partial tear ACL; Stump preserved ACL surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stump Preserving ACL Surgery (Experimental): Patients of partial tear ACL injury fulfilling inclusion criteria received stump preserving ACL surgery, entered conventional ACL reconstruction rehabilitation program
  Interventions: Other: conventional ACL rehabilitation program
- ACL Reconstruction (Active Comparator): Patients with complete tear ACL injury received ACL reconstruction entered conventional ACL rehabilitation program
  Interventions: Other: conventional ACL rehabilitation program

INTERVENTIONS:
Other: conventional ACL rehabilitation program — Conventional post-operative physical therapy exercises and rehabilitation, designed for ACL reconstruction for 6 months to 9 months.

SUMMARY:
Anterior cruciate ligament (ACL) is known to serve a number of functions in the knee joint. Besides providing mechanical stability, it also contributes to proprioceptive function. Numerous studies reported ACL is rich in mechanoreceptors contribute in proprioceptive function. ACL augmentation, or selective ACL bundle (AM, anteromedial or PL, posterolateral) reconstruction, a relatively new technique for partial torn ACL, preserves and augments the ACL remnant aiming at maintaining or facilitating proprioception, is now gaining its popularity. Preserving ACL stump is also reported to have merits in providing better mechanical protection and promoting revascularization to the newly reconstructed graft.

In local setting, stump preserving ACL surgery is the usual practice in handling partial ACL tear. With the background of the surgery's potential benefits in restoration of knee function, a single-blinded, comparative study on the difference in proprioception, postural stability and clinical outcome between stump preserving ACL surgery and reconstruction is conducted.

DETAILED DESCRIPTION:
Anterior cruciate ligament (ACL) is well known to be the knee's primary stabilizer which would be compromised by ligamentous injury, causing various functional deficits. Currently, ACL reconstruction is the common management focus on restoration of stability. Beside joint stabilization, proprioception, defined as the system of joint position sense and movement, is another function of the ACL which has also been widely studied.

The proprioceptive function of human ACL has been recognized since the 1980's. The first study by described the presence of mechanoreceptors in human ACL fibres. Study further proved that ACL is extensively innervated with neural elements.

Numerous studies reported ACL is rich in mechanoreceptors which contribute in proprioceptive function. One study on 29 ACL remnant reported that there are mechanoreceptors including Ruffini, Pacini receptors, Golgi tendon organ-like receptors and free nerves endings in the remnant and showed the numbers of mechanoreceptors is significantly related to joint sense accuracy. Another study performed by same group of researchers reported that a somatosensory evoked potential could be recorded in ACL remnants after electrical stimulation, confirmed original sensory neurons are preserved to certain extent, which may help graft neuralization and restoration of knee function. This further echos with various studies that, in ACL-deficit knee, loss of proprioceptive function is reported with corelation to the number of mechanoreceptors. At a result, it comes up with an idea that preserving the ACL remnant should help maintaining or facilitating proprioceptive function, by the operation technique of ACL augmentation.

ACL augmentation is a relatively new technique which preserves and augments the ACL remnant using extra graft. Under arthroscopic examination, if any of the ACL bundles, anteromedial (AM) and posterolateral (PL), shows a partial tear remnant of reasonable size, thickness and tension, augmentation may be performed instead of reconstruct the whole ligament. Instead of removing the remaining stump, it would be preserved as much as possible, and a formal ACL reconstruction would be performed. A commonly used graft is single-bundle autogenous semitendinosus gracilis tendon. As the retaining ACL fiber contains mechanoreceptor responsible for proprioception, it is believed that better knee proprioception and postural sense could be achieved by preserving the ACL remnant. Also, better vascularization and stronger mechanical protection is expected as native ACL fiber is retained.

The current management of partial tear ACL injury are mainly conservative treatment and surgical treatment, including reconstruction and augmentation. For augmentation, the common practise is to perform a "Selective Bundle Reconstruction", that is to reconstruct the torn bundle, either AM or PL reconstruction, and preserve the remaining intact one.

The clinical benefits of ACL augmentation had been reported by several studies. A study had demonstrated good clinical results in International Knee Documentation Commitee (IKDC) knee evaluation score, Cincinnati Knee Score and KT1000 in augmentation using autologous doubled and tripled semitendinosus (selective AM or PL) reconstruction at 1 year post-operatively.

An other comparison study between ACL augmentation (selective AM or PL reconstruction) and reconstruction showed superior result in knee anterior stability in clinical tests, KT2000 and knee joint position sense in augmentation group at a 2-year follow-up period. This study has demonstrated the post-operation comparison only and allogenic fascia lata graft was also used in the control reconstruction group, which is not a common graft to be used in ACL surgery in local setting. Moreover, as the assessment is performed at 2 years post-operatively, the more immediate and early post-operative effect of this surgical technique is still questionable.

As mentioned above, ACL augmentation may has potential clinical advantages including better knee stability, mechanical strength and proprioceptive function, yet evidence of the earlier effect of this technique is still lacking, with joint position sense was demonstrated by one study only. With the relatively new technique's popularity and potential benefit on proprioception, it deserves more research on studying the difference in both the clinical and proprioception outcome from reconstruction. Therefore, a comparative study on the difference in knee proprioception and postural stability between ACL augmentation and reconstruction, including early post-operative assessment is performed.

In local setting, if the ACL injury is noted to be partially torn from pre-operative Magnetic Resonance Imaging (MRI), surgeons would try to preserve the remaining stump as much as possible with a single bundle ACL reconstruction performed intra-operatively. In order to make the current study result meaningful and could be generalized in local setting, ACL augmentation is renamed as ACL stump-preserving surgery, which is the common practice in local setting.

ELIGIBILITY:
Inclusion Criteria:

* for stump reserving group: partial tear ACL injury with remnant of sizable, reasonable thickness and tension suitable
* for ACL reconstruction group: complete tear ACL injury
* for both groups: no complication such as wound infection after operation
* no history of medical problems, for example, heart disease

Exclusion Criteria:

* concomitant Medial Collateral Ligament (MCL), Lateral Collateral Ligament (LCL), Posterior Cruciate Ligament (PCL) injury, meniscus tear on the relevant knee
* previous or concomitant surgery on the relevant knee and other joints
* surgery or traumatic injuries to the contralateral limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-12 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Joint Position Sense 1 | Joint position sense at an expected average of 4 weeks before operation
  Using Biodex Dynamometer (Biodex Medical Systems, Shirley, NY, USA) for measurement.
Joint Position Sense 2 | Joint position sense at 1 month post-operation
  Using Biodex Dynamometer (Biodex Medical Systems, Shirley, NY, USA) for measurement.
Joint Position Sense 3 | Joint position sense at 3 month post-operation
  Using Biodex Dynamometer (Biodex Medical Systems, Shirley, NY, USA) for measurement.
Joint Position Sense 4 | Joint Position Sense at 6 months post-operation
  Using Biodex Dynamometer (Biodex Medical Systems, Shirley, NY, USA) for measurement.
Joint Position Sense 5 | Joint position sense at 1 year post-operation
  Using Biodex Dynamometer (Biodex Medical Systems, Shirley, NY, USA) for measurement.
Postural Balance 1 | Postural balance at an expected average of 4 weeks before operation
  Using Biodex Stability System (BSS; Biodex Medical Systems, Shirley, NY, USA with software version 3.1) for measurement
Postural Balance 2 | Postural balance at 1 month post-operation
  Using Biodex Stability System (BSS; Biodex Medical Systems, Shirley, NY, USA with software version 3.1) for measurement
Postural Balance 3 | Postural balance at 3 month post-operation
  Using Biodex Stability System (BSS; Biodex Medical Systems, Shirley, NY, USA with software version 3.1) for measurement
Postural Balance 4 | Postural balance at 6 month post-operation
  Using Biodex Stability System (BSS; Biodex Medical Systems, Shirley, NY, USA with software version 3.1) for measurement
Postural Balance 5 | Postural balance at 1 year post-operation
  Using Biodex Stability System (BSS; Biodex Medical Systems, Shirley, NY, USA with software version 3.1) for measurement

SECONDARY OUTCOMES:
Clinical Test 1 | Test at an expected average of 4 weeks before operation
  Anterior Drawer Test, Lachman Test and Knee range of motion
Clinical Test 2 | Post-operative 3 month
  Anterior Drawer Test, Lachman Test and Knee range of motion
Clinical Tests 3 | Post-operative 6 month
  Anterior Drawer Test, Lachman Test and Knee range of motion
Clinical Tests 4 | Post-operative 1 year
  Anterior Drawer Test, Lachman Test and Knee range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Holly KH Leung, Principal Investigator — Physiotherapy Department, Prince of Wales Hospital, Shatin, Hong Kong
Locations (1):
- Physiotherapy Department, Prince of Wales Hospital, Shatin, Hong Kong, China